CLINICAL TRIAL: NCT04377503
Title: Comparison of the Efficacy and Safety of Tocilizumab Versus Methylprednisolone in the Cytokine Release Syndrome of Patients With COVID-19. A Prospective Randomized Controlled Phase II Trial
Brief Title: Tocilizumab Versus Methylprednisolone in the Cytokine Release Syndrome of Patients With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The number of critically ill patients wirh COVID-19 decrease abruptly
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Principal investigator, Hospital Sao Domingos
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: covid-19 hsd
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2020-05

CONDITIONS: Cytokine Release Syndrome; Covid-19
Keywords: Cytokine release syndrome; COVID-19; Tocilizumab; Methylprednisolone; Safety; Efficacy
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19 | interventions — tocilizumab; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Patients will receive Tocilizumab, 8 mg / kg diluted in 100 ml of saline and administered IV for 60 minutes. The dose will be repeated only once 12 hours after the first dose.
  Interventions: Drug: Tocilizumab 180 MG/ML; Drug: Methylprednisolone Sodium Succinate
- Methylprednisolone (Active Comparator): Patients will receive methylprednisolone at a dose of 1.5 mg / kg / day divided into 2 daily doses for 7 days. Then they will receive 1 mg / kg / day for another 7 days in two daily doses. Finally 0.5 mg / kg / day for another 7 days.
  Interventions: Drug: Tocilizumab 180 MG/ML; Drug: Methylprednisolone Sodium Succinate

INTERVENTIONS:
Drug: Tocilizumab 180 MG/ML — Tocilizumab 8 mg/kg diluted in 100 ml of saline administered in 60 minutes. The dose will be repeated after 12 hours.
Drug: Methylprednisolone Sodium Succinate — Patients will receive methylprednisolone at a dose of 1.5 mg / kg / day divided into 2 daily doses for 7 days. Then they will receive 1 mg / kg / day for another 7 days. Finally 0.5 mg / kg / day until 21 days of use

SUMMARY:
This study compare the efficacy and safety of tocilizumab versus methylprednisolone in the cytokine release syndrome of patients with COVID-19

DETAILED DESCRIPTION:
In December 2019, several patients were diagnosed with pneumonia of undefined etiology in Wuhan, China. A few days later, a virus was identified as the etiologic agent. It was a new beta coronavirus that received the name of Severe Acute Respiratory Syndrome Coroinavirus (SARS-COV-2).

The disease quickly spread to the Wuhan region and in March reached northern Italy and soon across Europe. On March 14, the World Health Organization declared that COVID-19 had acquired seriousness and spread to be defined as a pandemic.

Since then, COVID-19 has challenged the ability of rich countries to meet the demand for beds, especially ICU beds, and it has also challenged science in search of effective treatment, while in record time research centers begins testing with a vaccine.

Although a significant percentage of patients with COVID-19 have a benign evolution, around 20% of cases the disease acquires sufficient severity from the point of view of lung involvement to justify treatment in the ICU. In addition, around 5% of patients evolve with extremely serious forms and are associated with a lethality of up to 60%. Some of these patients demonstrated in studies alterations in cellular and humoral immunity compatible with the cytokine release syndrome, an entity that has been described complicating the use of antineoplastic drugs and viral infections.

At this moment several studies, some of them with conclusions already seek to identify effective forms of treatment. Antiviral drugs such as Lopinavir-Ritonavir, which has already been tested in a prospective randomized study and has not been shown to be effective. The antiviral rendecivir was tested in a preliminary study brought a positive expectation and the hydroxychloroquine in studies with small samples is the drug that currently meets the highest expectations. None of these drugs, however, is effective in the case of the group of patients who acquire severity as a result of what has been called a cytokine storm. In this case, expectations are turned to interleukin antagonists and corticosteroids. Among the interleukin antagonists the drug that meets the most expectations is Tocilizumab, an interleukin-6 antagonist that has proven efficacy in the cytokine release syndrome caused by antineoplastic drugs. There are currently ongoing studies analyzing the role of tocilizumab and, at the same time, and along the same line, corticosteroids are being tested. There is currently no prospective randomized study examining the role of tocilizumab. Regarding corticosteroids, the only evidence comes from a retrospective study involving 201 patients with COVID pneumonia 19 and acute respiratory distress syndrome. This study showed an association between corticosteroids and reduced risk of death (HR 0.38; p = 0.003).

ELIGIBILITY:
Inclusion Criteria:

Men and non-pregnant women over 18 years old COVID diagnosis confirmed by real time polymerase chain reaction (RT-PCR) Pao2 / FIO2 <200 Laboratory: high sensitivity C reactive protein> 5 mg / L; lactic dehydrogenase (LDH ) > 245 U / l; Ferritin> 300; D-dimer> 1500; Interleukin-6> 7.0 pg / ml.

Exclusion Criteria:

* Known sensitivity/Allergy to tocilizumab
* Active tuberculosis
* Pregnancy
* Individuals, in the opinion of the investigators where progression to death is imminent and inevitable in the next 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Patient clinical status 15 days after randomization | 15 days after randomization
  A seven-category ordinal scale consisting of: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.

SECONDARY OUTCOMES:
Improving oxygenation | 15 days
  Improvement in PaO2/FIO2
Thorax CT improvement | 10 days
  Improvement in the computed tomography between D0 and D10 after randomization
ICU length of stay | 28 days
  Duration o ICU stay in days
Duration of mechanical ventilation | 28 days
  Days of mechanical ventilation
Incidence of acute kidney (AKI) with necessity of renal replacement therapy | 15 days
  AKI according to Kidney Disease Improving Global Outcomes (KDIGO)

CONTACTS AND LOCATIONS:
Overall Officials: PEDRO B FROTA, MD, Principal Investigator — Hospital Sao Domingos
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Ye Q, Wang B, Mao J. The pathogenesis and treatment of the ;Cytokine Storm' in COVID-19. J Infect. 2020 Jun;80(6):607-613. doi: 10.1016/j.jinf.2020.03.037. Epub 2020 Apr 10. PMID 32283152
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Grein J, Ohmagari N, Shin D, Diaz G, Asperges E, Castagna A, Feldt T, Green G, Green ML, Lescure FX, Nicastri E, Oda R, Yo K, Quiros-Roldan E, Studemeister A, Redinski J, Ahmed S, Bernett J, Chelliah D, Chen D, Chihara S, Cohen SH, Cunningham J, D'Arminio Monforte A, Ismail S, Kato H, Lapadula G, L'Her E, Maeno T, Majumder S, Massari M, Mora-Rillo M, Mutoh Y, Nguyen D, Verweij E, Zoufaly A, Osinusi AO, DeZure A, Zhao Y, Zhong L, Chokkalingam A, Elboudwarej E, Telep L, Timbs L, Henne I, Sellers S, Cao H, Tan SK, Winterbourne L, Desai P, Mera R, Gaggar A, Myers RP, Brainard DM, Childs R, Flanigan T. Compassionate Use of Remdesivir for Patients with Severe Covid-19. N Engl J Med. 2020 Jun 11;382(24):2327-2336. doi: 10.1056/NEJMoa2007016. Epub 2020 Apr 10. PMID 32275812
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524